CLINICAL TRIAL: NCT02779270
Title: Supervised Outdoor -Use Test for Sunscreen Products in Female Adults
Brief Title: Test the Outdoor Usage for Sunscreen Products in Female Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18318
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY987518 (Experimental): Subject will apply the test product to all sun exposed areas of face and body, wait for 15 minutes, then sunbathe for 30 minutes, exercise for 20 minutes, and then sunbathe for additional 30 minutes. Immediately after the second sunbathing, enter the pool and remain in the water for 20 minutes. Then repeat the sun and water exposure activities again.
  Interventions: Drug: BAY987518
- Sunscreen control (Active Comparator): Subject will apply the test product to all sun exposed areas of face and body, wait for 15 minutes, then sunbathe for 30 minutes, exercise for 20 minutes, and then sunbathe for additional 30 minutes. Immediately after the second sunbathing, enter the pool and remain in the water for 20 minutes. Then repeat the sun and water exposure activities again.
  Interventions: Drug: Sunscreen Lotion (U77-030 Control)

INTERVENTIONS:
Drug: BAY987518 — Apply the assigned test product to all sun-exposed areas of the face and body while avoiding contact with mouth, eyes and eyelids.
  Formulation: V27-104
  Arms: BAY987518
Drug: Sunscreen Lotion (U77-030 Control) — Apply the assigned test product to all sun-exposed areas of the face and body while avoiding contact with mouth, eyes and eyelids.
  Arms: Sunscreen control

SUMMARY:
To assess the safety of a sunscreen product when used outdoor.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy, fair skinned females between the ages of 18 to 65 years with no medical conditions of the skin.
* Subjects must have Fitzpatrick Skin Types I, II, III, or IV.
* Subjects must agree to restrict their sun exposure activities for at least five days.
* Subjects must be willing and physically able to spend approximately 3 continous hours in the sun.

Exclusion Criteria:

* Subjects must not have actinic keratoses, skin cancer, psoriasis, eczema, or any other acute or chronic skin conditions as determined by the dermatological medical history.
* Subjects must not have visible erythema, blistering, or peeling that would indicate recent sunburn.
* Subjects must not have significantly tanned skin.
* Subjects must not have received any phototoxic agent or any medication to which they have a known sensitivity or allergy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-09-26 (Actual); Primary Completion 2015-09-27 (Actual); Study Completion 2015-09-27 (Actual)

PRIMARY OUTCOMES:
Skin response to sun exposure according to the Skin Evaluation Response Scale from 0 to 3 | After approximately three hours direct sun-exposure

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States